CLINICAL TRIAL: NCT06516198
Title: A Pilot Study of the Utility of Auricular Acupressure in Enhancing Prehabilitation Benefits in Candidates for Thoracic Surgery.
Brief Title: Auricular Acupressure in Prehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB24-0888
Record Dates: First submitted 2024-06-12; First posted 2024-07-23 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Frailty; Thoracic; Prehabilitation; Lung Surgery; Wedge Resection; Segmentectomy; Lobectomy; Pneumonectomy; Status
Keywords: accupressure; vaccaria seeds
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant
Masking Description: A random number card will be drawn in sequence from a box. Even numbered cards will assign the patient to the experimental group, odd numbered cards will assign the patient to the control group. For the sham intervention (Sham Type II, same intervention with seeding and intermittent pressing) the seeds are placed at nonacupressure points for the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): A random number card will be drawn in sequence from a box. Even numbered cards will assign the patient to the experimental group, odd numbered cards will assign the patient to the control group.
  o Intervention group seed points:
  1. Shen Men (anxiety, depression, stress, pain)
  2. Point 0 (homeostasis, energy, mood)
  3. Endocrine (hormonal homeostasis)
  4. Subcortex (insomnia, anxiety, pain, inflammation)
  5. Autonomic (autonomic balance, pain)
  Interventions: Other: Auricular Acupressure
- Control Group (Sham Comparator): A random number card will be drawn in sequence from a box. Even numbered cards will assign the patient to the experimental group, odd numbered cards will assign the patient to the control group.
  o Control group sham seed points:
  1. Inside edge, center of tragus
  2. Helix midway between apex and tubercle
  3. Helix 1 cm anterior to apex
  4. 5 mm anterior to Shen Men
  5. Covered, 5 mm anterior and superior to endocrine
  For the sham intervention (Sham Type II, same intervention with seeding and intermittent pressing) the seeds are placed at nonacupressure points for the control group.
  Interventions: Other: Auricular Acupressure

INTERVENTIONS:
Other: Auricular Acupressure — Seeds will be placed during the clinic visit by the acupuncturist or the research associate according to the group the patient was assigned to. The care partner will observe the placement. A photograph of the seed placement will be taken and given to the care partner and to the patient after the relevant points are labeled by number or letter. The method of pressing is demonstrated for 1 one of the seeds, the care partner practices pressing on 2 other seeds, and the patient practices pressing on the remaining 2 seeds. Pressing consists of applying pressure, gradually increasing the pressure until the patient expresses discomfort, and maintaining that pressure until 2 minutes have passed. After pressing has been performed for each seed, the seeds are removed in clinic prior to clinic discharge.

SUMMARY:
Complementary medicine is recognized for its ability to enhance appetite, increase energy, reduce anxiety, decrease pain, and improve sleep, among many other benefits. Acupuncture is among the most frequent types of complementary medicine practiced in the US, and Medicare currently includes back pain as a reimbursable indication for this therapy. Acupuncture-related therapies may enhance efforts at prehabilitation in candidates for major lung resection.

DETAILED DESCRIPTION:
The plan is to use a small number of points for auricular acupressure that are selected to improve overall health, both physical and mental. Auricular acupuncture for management of pain using 5 points, informally referred to as "battlefield acupuncture" has demonstrated significant improvement in acute and chronic pain management. Auricular acupressure using a similarly small number of points has demonstrated improvement in chemotherapy-related disturbed sleep, fatigue, and appetite, postpartum depression and fatigue, and chemotherapy related fatigue and depression. It appears that auricular acupressure may be suitable for enhancing prehabilitation interventions for preoperative patients.

Patients will be selected from among individuals being considered for major lung surgery (wedge resection, segmentectomy, lobectomy, bilobectomy, or pneumonectomy; open or minimally invasive) who are expected to pursue a period of prehabilitation of 2 or more weeks prior to surgery.

ELIGIBILITY:
Inclusion Criteria

* Being considered for major lung surgery
* Surgery is not scheduled for at least 2 weeks
* Age ≥ 50 years
* Able to understand English at a 4th grade level
* No known contraindications to prehabilitation (strength, endurance, balance exercises)
* Able to provide informed consent for participation
* Has an adult care partner who will be available and capable of placing seeds
* Has access to smart phone for communication and image sharing
* Underwent frailty screening (given any score)
* Able to perform spirometry testing in clinic

Exclusion Criteria:

* Allergy to Vaccaria seeds
* Medical condition affecting either ear preventing use of auricular acupressure such as eczema, frostbite, sunburn

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-06-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled | 2 weeks
  The patient will complete a form after each seed pressing confirming the pressing and the time.

SECONDARY OUTCOMES:
Ease of participation in the study. | End of Study (Week 4)
  The patient will complete a form after each seed pressing confirming the pressing and the time.

OTHER OUTCOMES:
Accuracy of seed placement by a non-professional care partner. | Weekly until Week 4
  The care partner will place the seeds and then send a photo to the research team for correct seed placement verification or correction on a weekly basis. Accuracy of seed placement will be assessed by determining the number of corrections required to achieve seed placement each week.
The change of the intervention prehabilitation results | End of Study (Week 4)
  Compared to the control group, the intervention will demonstrate better increases in endurance, function, mood, breathing capacity, and strength.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lucia Madariaga, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang CS, Yang AW, Zhang AL, May BH, Xue CC. Sham control methods used in ear-acupuncture/ear-acupressure randomized controlled trials: a systematic review. J Altern Complement Med. 2014 Mar;20(3):147-61. doi: 10.1089/acm.2013.0238. Epub 2013 Oct 19. PMID 24138333
- [Result] Ferguson MK, Watson S, Johnson E, Vigneswaran WT. Predicted postoperative lung function is associated with all-cause long-term mortality after major lung resection for cancer. Eur J Cardiothorac Surg. 2014 Apr;45(4):660-4. doi: 10.1093/ejcts/ezt462. Epub 2013 Sep 19. PMID 24052607